CLINICAL TRIAL: NCT01653197
Title: Evive Health Randomized Controlled Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 813606-3
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: People Due for Mammogram; People Due for Colonoscopy; People Due for Blood Pressure Test; People Due for Cholesterol Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): On top of reminder, state: "Here's a fun fact to cheer you on your way:" and include a curiosity-inducing question and answer (e.g., "Q: Which is the only state that allows you to cast absentee ballots from outer space? // A: Texas")
  Interventions: Behavioral: Control
- Curiosity (Experimental): On top of reminder, state: "Here's a fun fact to cheer you on your way." and include a curiosity-inducing question (e.g., "Q: Which is the only state that allows you to cast absentee ballots from outer space?") Place the answer under a scratch-off patch ("A: Texas").
  Interventions: Behavioral: Curiosity
- Curiosity linked to Action (Experimental): On top of reminder, state: "Here's a fun fact to cheer you on your way. Reward yourself by scratching off the answer only after you've made your [colonoscopy/mammogram/etc.] appointment!" and include a curiosity-inducing question (e.g., "Q: Which is the only state that allows you to cast absentee ballots from outer space?") Place the answer under a scratch-off patch ("A: Texas")
  Interventions: Behavioral: Curiosity linked to Action

INTERVENTIONS:
Behavioral: Control — No scratch off element
  Arms: Control
Behavioral: Curiosity — The recipient will be prompted to scratch off for answer to question.
  Arms: Curiosity
Behavioral: Curiosity linked to Action — The recipient will be prompted to scratch off for answer only after he/she makes an appointment.
  Arms: Curiosity linked to Action

SUMMARY:
The mailer will encourage those who are due for mammograms, colonoscopies, blood pressure or cholesterol tests to receive the appropriate test. This particular mailer will only be sent to Evive clients in need to the test in question. The research will examine differences in follow-through on this recommendation among the targeted population over the 3-12 month period following the mailing as a function of experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* Employee at partner corporation
* Due for mammogram, colonoscopy, blood pressure or cholesterol test

Exclusion Criteria:

* Already received mammogram, colonoscopy, blood pressure or cholesterol test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants who follow-through from the mailing | three to twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States